CLINICAL TRIAL: NCT04618549
Title: Direct Anterior Approach (in Regular OR Table) Versus Mini Posterior Approach Versus Lateral Approach for the Treatment of Displaced Femoral Neck Fractures: A Prospective Randomized Trial
Brief Title: Direct Anterior Approach Versus Mini Posterior Approach Versous Lateral Approach for Displaced Femoral Neck Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Vasileios S. Nikolaou, Associate Professor of Orthopaedics, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2020-06-17; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Hip Fractures; Femoral Neck Fractures
Keywords: hip; fractures; surgical approach; outcome; bleeding
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures; Fractures, Bone; Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Direct anterior approach (Active Comparator): Patients with a femoral neck fracture, treated by hemiarthroplasty by direct anterior approach, using a regular OR table, without hip hyperextension.
  Interventions: Procedure: Direct Anterior Approach Hemiarthroplasty
- Mini Posterior Approach (Active Comparator): Patients with a femoral neck fracture, treated by hemiarthroplasty by a mini posterior approach.
  Interventions: Procedure: Mini Posterior Approach
- Lateral approach (Active Comparator): Patients with a femoral neck fracture, treated by hemiarthroplasty by a lateral (Hardinge) approach.
  Interventions: Procedure: Lateral approach

INTERVENTIONS:
Procedure: Direct Anterior Approach Hemiarthroplasty — Hemiarthroplasty to elderly patients with femoral neck fracture through a direct anterior approach
  Arms: Direct anterior approach
Procedure: Mini Posterior Approach — Hemiarthroplasty to elderly patients with femoral neck fracture through a mini posterior approach
  Arms: Mini Posterior Approach
Procedure: Lateral approach — Hemiarthroplasty to elderly patients with femoral neck fracture through a lateral approach (Hardinge)
  Arms: Lateral approach

SUMMARY:
In general, hip fractures in the elderly are associated with a high one year-mortality up to 36 %. Apart from choosing the proper treatment, optimizing the surgical technique itself offers options to improve the outcome. Early mobilization after hip hemi¬arthroplasty correlates with improved ambulation, reduced need for assisted transfers, and less use of extended care facilities after hospital discharge.

Nowadays, in order to reduce soft tissue damage and gain quicker postoperative recovery and faster rehabilitation, various MIS techniques have been proposed. Two of these techniques are the mini posterior approach and the mini direct anterior approach. The direct anterior approach was developed as a true internervous and intermuscular surgical approach with proposed benefits of faster recovery, quicker return to function, and less pain. In theory, the direct anterior approach should cause less tissue damage than mini posterior approach, as it is performed through a plane between neurlogical tissue and intermuscular plane without muscle transection.

The aim of this study is to evaluate the clinical and radiological outcomes of the direct anterior approach for bipolar head endoprosthetic hemiarthroplasty in patients with displaced femoral neck fractures in comparison with the mini posterior approach and the traditional lateral approach, for the treatment of the same fractures. The investigators hypothesized that patients undergoing the direct anterior approach would have better clinical and radiological results in comparison with the mini posterior and lateral approach.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing hip fracture surgery for displaced femoral neck fractures (Garden 3 and 4 fractures) and treated by cemented hemiarthroplasty will be included in the study. Patients must have the ability to give informed consent or a legal guardian is available.

Exclusion Criteria:

* The exclusion criteria include open or pathological fractures, re-fractures, infection, concomitant injuries of the ipsi- or contralateral leg or upper limb, skin diseases in the area of proposed incisions, patients that are mentally incapable of understanding the consequences of the study and reduced compliance.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
The Five Item Barthel Index | 6 weeks post-surgery
  Patient mobilization and motoric status measured with a five-item-Barthel index.
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. The Barthel Index is a widely used measure of physical dependence in personal activities of daily living (PADL). The short five-item Barthel index score ranges from 0-15 points, with 0 means the worst score and 15 the optimal score that a patient can achieve.
The Five Item Barthel Index | 3 months post-surgery
  Patient mobilization and motoric status measured with a five-item-Barthel index.
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. The Barthel Index is a widely used measure of physical dependence in personal activities of daily living (PADL). The short five-item Barthel index score ranges from 0-15 points, with 0 means the worst score and 15 the optimal score that a patient can achieve.
The Timed Up and Go test (TUG) | 4 days after the surgery
  The Timed Up and Go test, is a test of balance that is commonly used to examine functional mobility in community-dwelling, frail older adults. The test requires a subject to stand up, walk 3 m (10 ft), turn, walk back, and sit down. Time taken to complete the test is strongly correlated to the level of functional mobility.
  Older adults who are able to complete the task in less than 20 seconds have been shown to be independent in transfer tasks involved in activities of daily living, and walk at gait speeds that should be sufficient for community mobility (0.5 m/s). In contrast, older adults requiring 30 seconds or longer to complete the task tend to be more dependent on activities of daily living and require assistive devices for ambulation.
The Timed Up and Go test (TUG) | 6 weeks post surgery
  The Timed Up and Go test, is a test of balance that is commonly used to examine functional mobility in community-dwelling, frail older adults. The test requires a subject to stand up, walk 3 m (10 ft), turn, walk back, and sit down. Time taken to complete the test is strongly correlated to the level of functional mobility.
  Older adults who are able to complete the task in less than 20 seconds have been shown to be independent in transfer tasks involved in activities of daily living, and walk at gait speeds that should be sufficient for community mobility (0.5 m/s). In contrast, older adults requiring 30 seconds or longer to complete the task tend to be more dependent on activities of daily living and require assistive devices for ambulation.
Parker mobility score | One week before the fracture occur
  Postoperative mobility score, as proposed by Parker and Palmer (Parker MJ, Palmer CR, JBJS Br (1993) ).
  The Parker Mobility Score is a composite measurement of the patient's mobility indoors, outdoors and during shopping, and is used in studies either to measure the mobility as an outcome measure or as a predictor for mortality
  Range 0-9 points (0 is the worst score and 9 the best score that a patient can achieve)
Parker mobility score | 3 months post surgery
  Postoperative mobility score, as proposed by Parker and Palmer (Parker MJ, Palmer CR, JBJS Br (1993) ).
  The Parker Mobility Score is a composite measurement of the patient's mobility indoors, outdoors and during shopping, and is used in studies either to measure the mobility as an outcome measure or as a predictor for mortality
  Range 0-9 points (0 is the worst score and 9 the best score that a patient can achieve)

SECONDARY OUTCOMES:
Change to the Total blood loss (TBL) | Preop to day 4 post surgery
  For calculation of the total blood loss (TBL) expressed to total Hb loss and total Volume loss , we will use the number of transfusions (55 grams of haemoglobin per transfusion), the haemoglobin concentration on preoperatively (Hgbi) and the haemoglobin concentration on the last available measure of haemoglobin concentration (Hgbe). (Hemoglobin balance method)
Change at the Pain Visual Analog (VAS) score | From day one up to 6 weeks post surgery
  The pain visual analog scale (VAS) is commonly used as the outcome measure for pain. It is presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" (0 pain) and "worst pain imaginable." (100 pain)
Muscle Damage Markers | Daily for days 1-4 Post-op
  CK (Creatine Kinase), ECR and CRP
Change at Creatine Kinase (CK) | Daily for days 1-4 Post-op and at 6 weeks post-op
  The appearance of creatine kinase (CK) in blood has been generally considered to be an indirect marker of muscle damage.
  Reference Values Males >3 months: 39-308 U/L Females >3 months: 26-192 U/L
Change at C-Reactive protein (CRP) | Daily for days 1-4 Post-op and at 6 weeks post-op
  C-reactive protein (CRP) levels have been documented as a potent marker for skeletal muscle damage.
  Reference Value: 0-10mg/L